CLINICAL TRIAL: NCT06837181
Title: Studying the Presence of CFRD Complications With Thoughtful Recruitment (SPeCTRuM)
Acronym: SPeCTRuM
Status: Recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SPeCTRuM; 007365A124 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2025-01-29; First posted 2025-02-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis-related Diabetes; Diabetes; Retinopathy; Neuropathy; Nephropathy; Blood Pressure; Cardiovascular Risk; Microvascular
Keywords: Cystic Fibrosis; CFRD; Cystic Fibrosis-Related Diabetes; Observational; Physical Activity Tracker; Continuous glucose monitoring; CGM; Diabetes; blood pressure; cardiovascular risk; microvascular; diabetes complications; social determinants of health
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus; Retinal Diseases; Kidney Diseases; Diabetes Complications | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Cystic Fibrosis-Related Diabetes: Individuals diagnosed with Cystic Fibrosis-Related Diabetes for more than 5 years before enrollment
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — This is an observational study.

SUMMARY:
This multicenter cross-sectional study will include a diverse population of adolescents and adults with CF.

The overall Aim is to describe prevalence of diabetes microvascular complications and macrovascular surrogates in people with established CFRD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable) obtained from participant or participant's legally authorized representative
* For Adults: Must be able to consent on one own's behalf (i.e., cannot lack cognitive capacity to consent due to the required patient-reported outcomes)
* Be willing and able to adhere to the study protocol requirements
* Age ≥ 12 years at time of enrollment
* CF diagnosis based on two CF causing mutations and/or positive sweat test according to CFF diagnostic criteria
* CFRD diagnosis ≥ 5 years at time of enrollment

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk to the subject
* History of transplant
* Pregnancy reported by participant at time of consent or at any point during active study participation

Pulse Wave Velocity Exclusion Criteria:

* Erratic, accelerated or mechanically controlled irregular heart rhythms including arrhythmias
* Carotid or aortic valve stenosis
* Peripheral artery disease or leg artery disease
* Generalized constriction or localized spasm of muscular conduit arteries such as seen immediately after hypothermic cardiopulmonary bypass surgery or accompanying Raynaud's phenomena or intense cold.
* Possible exclusions based on investigator medical provider assessment (additional precautions may be followed to allow inclusion):

  * Pressure reading should not be conducted on a limb where there is intravenous access, arterio-venous shunt, or where circulation is compromised.
  * Pressure reading should not be conducted on the side of the body that a mastectomy was done.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with CFRD diagnosis ≥ 5 years at time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular Complications | From enrollment to the end of the participant's participation or 4 weeks
  To describe the rates of microvascular complications (retinopathy, nephropathy, and peripheral neuropathy) and their relationships with HbA1c and diabetes duration in diverse cohort of adolescents and adults with CFRD for ≥5 years.
Macrovascular Surrogates | From enrollment to the end of the participant's participation or 4 weeks
  To describe macrovascular surrogates (resting blood pressure (BP), fasting lipids) and their relationship with HbA1c, diabetes duration and BMI in a diverse cohort with established CFRD.

SECONDARY OUTCOMES:
PhenX English Proficiency | From enrollment to the end of the participant's participation or 4 weeks
  This questionnaire will be used to describe the social determinants of health in the study population and their cross-sectional relationships with microvascular complications and macrovascular surrogates will largely be explored.
PhenX Food Security & Prescription Accessibility | From enrollment to the end of the participant's participation or 4 weeks
  This questionnaire will be used to describe the social determinants of health in the study population and their cross-sectional relationships with microvascular complications and macrovascular surrogates will largely be explored.
Exercise and Substance Use | From enrollment to the end of the participant's participation or 4 weeks
  This questionnaire ask questions regarding participants' physical activity, sleeping habits and substance use.
Pubertal Self-Assessment | From enrollment to the end of the participant's participation or 4 weeks
  A self-evaluation questionnaire to assess child's pubertal development.
Beverage Questionnaire (BEVQ15) | From enrollment to the end of the participant's participation or 4 weeks
  A questionnaire that asks the frequency and amount of beverage intake for the past month.
CFRD Care & Technology | From enrollment to the end of the participant's participation or 4 weeks
  This is a questionnaire that asks participants regarding their CFRD care and the technology they use to help them manage diabetes.
Diabetes Management Experience | From enrollment to the end of the participant's participation or 4 weeks
  This is a questionnaire that asks how participants manage their diabetes for the past 12 months.
Problem Areas in Diabetes (PAID) | From enrollment to the end of the participant's participation or 4 weeks
  Questionnaire that asks participants about possible diabetes-related issues they have experienced.
Problem Areas in Diabetes Parents of Teens (P-PAID-T) | From enrollment to the end of the participant's participation or 4 weeks
  Questionnaire about what the parent or guardian of a participant may experience with their child's diabetes and rating how true it is for them over the past month.
Hypoglycemia Fear Survey (Child) | From enrollment to the end of the participant's participation or 4 weeks
  A survey that consists of 25 questions and selecting from scale (0 = never to 4 = always) about how low blood sugar makes children feel and do.
Hypoglycemia Fear Survey (Parent) | From enrollment to the end of the participant's participation or 4 weeks
  Survey that consists of 25 questions about the frequency of things parents of children with diabetes sometimes do to keep from having low blood sugar.
Hypoglycemia Fear Survey (Adult-Short Form)/Worry (HFS-II-Worry) | From enrollment to the end of the participant's participation or 4 weeks
  A survey about various scenarios that may happen to the participant and rating how true it is for them over the past 6 months.
Gold Score | From enrollment to the end of the participant's participation or 4 weeks
  A 7 item scale that measures hypoglycemia awareness
All of Us | From enrollment to the end of the participant's participation or 4 weeks
  A questionnaire that consists of 14 questions asking about the participant, their work and their home life.
Continuous glucose monitoring (CGM)-defined glycemic control (time-in-range, time-above-range, time-below-range, glucose variability), and the relationships between CGM metrics and HbA1c, in a diverse population of people with established CFRD | 3-10 days
  This will be measured using a continuous glucose monitor that will be worn by the participant for 3 to 10 days.
Diversity of participants enrolled and barriers to enrollment | From enrollment to the end of the participant's participation or 4 weeks
  This will be measured using the patient-related outcomes questionnaires.
Renal function by eGFR | From enrollment to the end of the participant's participation or 4 weeks
  Function will be assessed by collection of creatinine and Cystatin-C
Liver function | From enrollment to the end of the participant's participation or 4 weeks
  This will be measured by liver enzymes and complete blood count (CBC); APRI and EMR data for liver imaging

OTHER OUTCOMES:
Exploratory Outcome - Participant diversity | From enrollment to the end of the participant's participation or 4 weeks
  This will measure diversity of individuals who were approached for study inclusion, who were recruited, who consented and who partially or fully completed study procedures as well as barriers and facilitators to recruitment.
Cardiovascular sub-study - Pulse Wave Velocity and Pulse Wave Analysis (PWV & PWA) | 1 study visit day
  A Sphygmocor XCEL device will be used to measure PWV/PWA (m/sec), pulse pressure amplification and augmentation index (Aix) and Aix adjusted to a HR of 75 (Aix-75).
Exploratory Outcome - HbA1c and CGM metrics with nutritional intake | 3 days
  The participant will complete 3-day recall of food intake using NIH's Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool.
Exploratory Outcome - HbA1c and CGM metrics with physical activity | 3-10 days
  The participant will be required to wear an accelerometer device for 3 to 10 days to assess physical activity.
Cardiovascular sub-study - Ambulatory Blood Pressure Monitoring | 24 hours
  An oscillometric Spacelab monitors will be used to measure variables including SBP/DBP and BP load (%BP above 95th percentile for sex and height) for the 24-hour period and awake/sleep period. Sleep time will be determined from actigraphy and participant documentation.
Fecal Collection | From enrollment to the end of the participant's participation or 4 weeks
  Participant stool sample will be obtained for fecal elastase only for those for pancreatic sufficiency status is unclear.
Sample Collection for Biorepository | From enrollment to the end of the participant's participation or 4 weeks
  Blood, urine and stool will be collected for biorepository.
Information Collection for Geocoding | from enrollment
  The study will use the participants' addresses or part of their addresses (such as their zip codes) to allow researchers to look at how where they live might be related to their health through geocoding.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Keck Medical Center of USC, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Massachusetts, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University Cystic Fibrosis Program, New York, New York
  - Atrium Health Wake Forest Baptist (Wake Forest Baptist), Winston-Salem, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charlestone, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agbaje AO, Barker AR, Tuomainen TP. Differing Relations Of Arterial Stiffness And Carotid Intima-Media Thickness In Adolescence With Metabolic Risks In Young Adulthood: The ALSPAC Study. Circulation. 2021;144(Suppl_1):A13236-A. doi: doi:10.1161/circ.144.suppl_1.13236
- [Background] Kelly A, Magge SN, Walega R, Cochrane C, Pipan ME, Zemel BS, Cohen MS, Gidding SS, Townsend R. Cross-Sectional Study of Arterial Stiffness in Adolescents with Down Syndrome. J Pediatr. 2019 Sep;212:79-86.e1. doi: 10.1016/j.jpeds.2019.04.059. Epub 2019 Jun 11. PMID 31201031
- [Background] DeLoach SS, Townsend RR. Vascular stiffness: its measurement and significance for epidemiologic and outcome studies. Clin J Am Soc Nephrol. 2008 Jan;3(1):184-92. doi: 10.2215/CJN.03340807. PMID 18178784
- [Background] Feldman EL, Stevens MJ, Thomas PK, Brown MB, Canal N, Greene DA. A practical two-step quantitative clinical and electrophysiological assessment for the diagnosis and staging of diabetic neuropathy. Diabetes Care. 1994 Nov;17(11):1281-9. doi: 10.2337/diacare.17.11.1281. PMID 7821168
- [Background] Bergman M, Tuomilehto J. International Diabetes Federation Position Statement on the 1-hour post-load plasma glucose for the diagnosis of intermediate hyperglycaemia and type 2 diabetes. Diabetes Res Clin Pract. 2024 Apr;210:111636. doi: 10.1016/j.diabres.2024.111636. Epub 2024 Mar 25. No abstract available. PMID 38537890
- [Background] Bergman M, Manco M, Satman I, Chan J, Schmidt MI, Sesti G, Vanessa Fiorentino T, Abdul-Ghani M, Jagannathan R, Kumar Thyparambil Aravindakshan P, Gabriel R, Mohan V, Buysschaert M, Bennakhi A, Pascal Kengne A, Dorcely B, Nilsson PM, Tuomi T, Battelino T, Hussain A, Ceriello A, Tuomilehto J. International Diabetes Federation Position Statement on the 1-hour post-load plasma glucose for the diagnosis of intermediate hyperglycaemia and type 2 diabetes. Diabetes Res Clin Pract. 2024 Mar;209:111589. doi: 10.1016/j.diabres.2024.111589. Epub 2024 Mar 7. PMID 38458916
- [Background] McGarry M. Transparency and diversity in cystic fibrosis research. Lancet. 2020 Aug 29;396(10251):601. doi: 10.1016/S0140-6736(20)30906-5. No abstract available. PMID 32861304
- [Background] Kartal Ozturk G, Conkar S, Eski A, Gulen F, Keskinoglu A, Demir E. Evaluation of increased arterial stiffness in pediatric patients with cystic fibrosis by augmentation index and pulse wave velocity analysis. Pediatr Pulmonol. 2020 May;55(5):1147-1153. doi: 10.1002/ppul.24688. Epub 2020 Feb 14. PMID 32057197
- [Background] Eising JB, van der Ent CK, Teske AJ, Vanderschuren MM, Uiterwaal CSPM, Meijboom FJ. Young patients with cystic fibrosis demonstrate subtle alterations of the cardiovascular system. J Cyst Fibros. 2018 Sep;17(5):643-649. doi: 10.1016/j.jcf.2017.12.009. Epub 2018 Feb 3. PMID 29398489
- [Background] Buehler T, Steinmann M, Singer F, Regamey N, Casaulta C, Schoeni MH, Simonetti GD. Increased arterial stiffness in children with cystic fibrosis. Eur Respir J. 2012 Jun;39(6):1536-7. doi: 10.1183/09031936.00212511. No abstract available. PMID 22654008
- [Background] Urbina EM, Isom S, Bell RA, Bowlby DA, D'Agostino R Jr, Daniels SR, Dolan LM, Imperatore G, Marcovina SM, Merchant AT, Reynolds K, Shah AS, Wadwa RP, Dabelea D; SEARCH for Diabetes in Youth Study Group. Burden of Cardiovascular Risk Factors Over Time and Arterial Stiffness in Youth With Type 1 Diabetes Mellitus: The SEARCH for Diabetes in Youth Study. J Am Heart Assoc. 2019 Jul 2;8(13):e010150. doi: 10.1161/JAHA.118.010150. Epub 2019 Jun 19. PMID 31213111
- [Background] Stoner L, Kucharska-Newton A, Meyer ML. Cardiometabolic Health and Carotid-Femoral Pulse Wave Velocity in Children: A Systematic Review and Meta-Regression. J Pediatr. 2020 Mar;218:98-105.e3. doi: 10.1016/j.jpeds.2019.10.065. Epub 2019 Dec 4. PMID 31810627
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] Mendizabal B, Urbina EM. Subclinical Atherosclerosis in Youth: Relation to Obesity, Insulin Resistance, and Polycystic Ovary Syndrome. J Pediatr. 2017 Nov;190:14-20. doi: 10.1016/j.jpeds.2017.06.043. Epub 2017 Jul 13. No abstract available. PMID 28712518
- [Background] Khoury M, Urbina EM. Hypertension in adolescents: diagnosis, treatment, and implications. Lancet Child Adolesc Health. 2021 May;5(5):357-366. doi: 10.1016/S2352-4642(20)30344-8. Epub 2021 Mar 10. PMID 33711291
- [Background] Cote AT, Phillips AA, Harris KC, Sandor GG, Panagiotopoulos C, Devlin AM. Obesity and arterial stiffness in children: systematic review and meta-analysis. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):1038-44. doi: 10.1161/ATVBAHA.114.305062. Epub 2015 Jan 29. PMID 25633314
- [Background] Agbaje AO, Barker AR, Tuomainen TP. Effects of Arterial Stiffness and Carotid Intima-Media Thickness Progression on the Risk of Overweight/Obesity and Elevated Blood Pressure/Hypertension: a Cross-Lagged Cohort Study. Hypertension. 2022 Jan;79(1):159-169. doi: 10.1161/HYPERTENSIONAHA.121.18449. Epub 2021 Nov 17. PMID 34784721
- [Background] Agbaje AO, Barker AR, Tuomainen TP. Cardiorespiratory Fitness, Fat Mass, and Cardiometabolic Health with Endothelial Function, Arterial Elasticity, and Stiffness. Med Sci Sports Exerc. 2022 Jan 1;54(1):141-152. doi: 10.1249/MSS.0000000000002757. PMID 34334718
- [Background] Agbaje AO, Barker AR, Mitchell GF, Tuomainen TP. Effect of Arterial Stiffness and Carotid Intima-Media Thickness Progression on the Risk of Dysglycemia, Insulin Resistance, and Dyslipidemia: a Temporal Causal Longitudinal Study. Hypertension. 2022 Mar;79(3):667-678. doi: 10.1161/HYPERTENSIONAHA.121.18754. Epub 2022 Jan 18. PMID 35038890
- [Background] Townsend RR, Wilkinson IB, Schiffrin EL, Avolio AP, Chirinos JA, Cockcroft JR, Heffernan KS, Lakatta EG, McEniery CM, Mitchell GF, Najjar SS, Nichols WW, Urbina EM, Weber T; American Heart Association Council on Hypertension. Recommendations for Improving and Standardizing Vascular Research on Arterial Stiffness: A Scientific Statement From the American Heart Association. Hypertension. 2015 Sep;66(3):698-722. doi: 10.1161/HYP.0000000000000033. Epub 2015 Jul 9. No abstract available. PMID 26160955
- [Background] Mitchell GF. Arterial Stiffness in Aging: Does It Have a Place in Clinical Practice?: Recent Advances in Hypertension. Hypertension. 2021 Mar 3;77(3):768-780. doi: 10.1161/HYPERTENSIONAHA.120.14515. Epub 2021 Feb 1. PMID 33517682
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Chirinos JA, Segers P, Hughes T, Townsend R. Large-Artery Stiffness in Health and Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Sep 3;74(9):1237-1263. doi: 10.1016/j.jacc.2019.07.012. PMID 31466622
- [Background] Boutouyrie P, Chowienczyk P, Humphrey JD, Mitchell GF. Arterial Stiffness and Cardiovascular Risk in Hypertension. Circ Res. 2021 Apr 2;128(7):864-886. doi: 10.1161/CIRCRESAHA.121.318061. Epub 2021 Apr 1. PMID 33793325
- [Background] Karnsakul W, Wasuwanich P, Ingviya T, Vasilescu A, Carson KA, Mogayzel PJ, Schwarz KB. A longitudinal assessment of non-invasive biomarkers to diagnose and predict cystic fibrosis-associated liver disease. J Cyst Fibros. 2020 Jul;19(4):546-552. doi: 10.1016/j.jcf.2020.05.002. Epub 2020 May 30. PMID 32482593
- [Background] Ayoub F, Trillo-Alvarez C, Morelli G, Lascano J. Risk factors for hepatic steatosis in adults with cystic fibrosis: Similarities to non-alcoholic fatty liver disease. World J Hepatol. 2018 Jan 27;10(1):34-40. doi: 10.4254/wjh.v10.i1.34. PMID 29399276
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Khosla L, Bhat S, Fullington LA, Horlyck-Romanovsky MF. HbA1c Performance in African Descent Populations in the United States With Normal Glucose Tolerance, Prediabetes, or Diabetes: A Scoping Review. Prev Chronic Dis. 2021 Mar 11;18:E22. doi: 10.5888/pcd18.200365. PMID 33705304
- [Background] Herman WH. Are There Clinical Implications of Racial Differences in HbA1c? Yes, to Not Consider Can Do Great Harm! Diabetes Care. 2016 Aug;39(8):1458-61. doi: 10.2337/dc15-2686. PMID 27457636
- [Background] Yapanis M, James S, Craig ME, O'Neal D, Ekinci EI. Complications of Diabetes and Metrics of Glycemic Management Derived From Continuous Glucose Monitoring. J Clin Endocrinol Metab. 2022 May 17;107(6):e2221-e2236. doi: 10.1210/clinem/dgac034. PMID 35094087
- [Background] Xu Y, Bergenstal RM, Dunn TC, Ram Y, Ajjan RA. Interindividual variability in average glucose-glycated haemoglobin relationship in type 1 diabetes and implications for clinical practice. Diabetes Obes Metab. 2022 Sep;24(9):1779-1787. doi: 10.1111/dom.14763. Epub 2022 Jun 2. PMID 35546274
- [Background] Scully KJ, Sherwood JS, Martin K, Ruazol M, Marchetti P, Larkin M, Zheng H, Sawicki GS, Uluer A, Neuringer I, Yonker LM, Sicilian L, Wexler DJ, Putman MS. Continuous Glucose Monitoring and HbA1c in Cystic Fibrosis: Clinical Correlations and Implications for CFRD Diagnosis. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1444-e1454. doi: 10.1210/clinem/dgab857. PMID 34850006
- [Background] Chan CL, Steck AK, Severn C, Pyle L, Rewers M, Zeitler PS. Lessons From Continuous Glucose Monitoring in Youth With Pre-Type 1 Diabetes, Obesity, and Cystic Fibrosis. Diabetes Care. 2020 Mar;43(3):e35-e37. doi: 10.2337/dc19-1690. Epub 2020 Jan 14. No abstract available. PMID 31937609
- [Background] Chan CL, Pyle L, Vigers T, Zeitler PS, Nadeau KJ. The Relationship Between Continuous Glucose Monitoring and OGTT in Youth and Young Adults With Cystic Fibrosis. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e548-e560. doi: 10.1210/clinem/dgab692. PMID 34537845
- [Background] O'Riordan SM, Hindmarsh P, Hill NR, Matthews DR, George S, Greally P, Canny G, Slattery D, Murphy N, Roche E, Costigan C, Hoey H. Validation of continuous glucose monitoring in children and adolescents with cystic fibrosis: a prospective cohort study. Diabetes Care. 2009 Jun;32(6):1020-2. doi: 10.2337/dc08-1925. Epub 2009 Mar 11. PMID 19279304
- [Background] Shoemaker MJ, Hurt H, Arndt L. The evidence regarding exercise training in the management of cystic fibrosis: a systematic review. Cardiopulm Phys Ther J. 2008 Sep;19(3):75-83. PMID 20467502
- [Background] Dwyer TJ, Elkins MR, Bye PT. The role of exercise in maintaining health in cystic fibrosis. Curr Opin Pulm Med. 2011 Nov;17(6):455-60. doi: 10.1097/MCP.0b013e32834b6af4. PMID 21881514
- [Background] Beaudoin N, Bouvet GF, Coriati A, Rabasa-Lhoret R, Berthiaume Y. Combined Exercise Training Improves Glycemic Control in Adult with Cystic Fibrosis. Med Sci Sports Exerc. 2017 Feb;49(2):231-237. doi: 10.1249/MSS.0000000000001104. PMID 27669451
- [Background] Hamilton CM, Strader LC, Pratt JG, Maiese D, Hendershot T, Kwok RK, Hammond JA, Huggins W, Jackman D, Pan H, Nettles DS, Beaty TH, Farrer LA, Kraft P, Marazita ML, Ordovas JM, Pato CN, Spitz MR, Wagener D, Williams M, Junkins HA, Harlan WR, Ramos EM, Haines J. The PhenX Toolkit: get the most from your measures. Am J Epidemiol. 2011 Aug 1;174(3):253-60. doi: 10.1093/aje/kwr193. Epub 2011 Jul 11. PMID 21749974
- [Background] Petersen MC, Begnel L, Wallendorf M, Litvin M. Effect of elexacaftor-tezacaftor-ivacaftor on body weight and metabolic parameters in adults with cystic fibrosis. J Cyst Fibros. 2022 Mar;21(2):265-271. doi: 10.1016/j.jcf.2021.11.012. Epub 2021 Dec 1. PMID 34862121
- [Background] Gary-Webb TL, Suglia SF, Tehranifar P. Social epidemiology of diabetes and associated conditions. Curr Diab Rep. 2013 Dec;13(6):850-9. doi: 10.1007/s11892-013-0427-3. PMID 24085624
- [Background] Hill-Briggs F, Adler NE, Berkowitz SA, Chin MH, Gary-Webb TL, Navas-Acien A, Thornton PL, Haire-Joshu D. Social Determinants of Health and Diabetes: A Scientific Review. Diabetes Care. 2020 Nov 2;44(1):258-79. doi: 10.2337/dci20-0053. Online ahead of print. No abstract available. PMID 33139407
- [Background] Haire-Joshu D, Hill-Briggs F. The Next Generation of Diabetes Translation: A Path to Health Equity. Annu Rev Public Health. 2019 Apr 1;40:391-410. doi: 10.1146/annurev-publhealth-040218-044158. Epub 2019 Jan 2. PMID 30601723
- [Background] Haw JS, Shah M, Turbow S, Egeolu M, Umpierrez G. Diabetes Complications in Racial and Ethnic Minority Populations in the USA. Curr Diab Rep. 2021 Jan 9;21(1):2. doi: 10.1007/s11892-020-01369-x. PMID 33420878
- [Background] Lado JJ, Lipman TH. Racial and Ethnic Disparities in the Incidence, Treatment, and Outcomes of Youth with Type 1 Diabetes. Endocrinol Metab Clin North Am. 2016 Jun;45(2):453-61. doi: 10.1016/j.ecl.2016.01.002. Epub 2016 Apr 7. PMID 27241975
- [Background] Walker AF, Schatz DA, Johnson C, Silverstein JH, Rohrs HJ. Disparities in social support systems for youths with type 1 diabetes. Clin Diabetes. 2015 Apr;33(2):62-9. doi: 10.2337/diaclin.33.2.62. PMID 25897185
- [Background] Centers for Disease Control and Prevention (CDC). Racial disparities in diabetes mortality among persons aged 1-19 years--United States, 1979-2004. MMWR Morb Mortal Wkly Rep. 2007 Nov 16;56(45):1184-7. PMID 18004236
- [Background] Willi SM, Miller KM, DiMeglio LA, Klingensmith GJ, Simmons JH, Tamborlane WV, Nadeau KJ, Kittelsrud JM, Huckfeldt P, Beck RW, Lipman TH; T1D Exchange Clinic Network. Racial-ethnic disparities in management and outcomes among children with type 1 diabetes. Pediatrics. 2015 Mar;135(3):424-34. doi: 10.1542/peds.2014-1774. PMID 25687140
- [Background] Valenzuela JM, Seid M, Waitzfelder B, Anderson AM, Beavers DP, Dabelea DM, Dolan LM, Imperatore G, Marcovina S, Reynolds K, Yi-Frazier J, Mayer-Davis EJ; SEARCH for Diabetes in Youth Study Group. Prevalence of and disparities in barriers to care experienced by youth with type 1 diabetes. J Pediatr. 2014 Jun;164(6):1369-75.e1. doi: 10.1016/j.jpeds.2014.01.035. Epub 2014 Feb 25. PMID 24582008
- [Background] Kahkoska AR, Shay CM, Crandell J, Dabelea D, Imperatore G, Lawrence JM, Liese AD, Pihoker C, Reboussin BA, Agarwal S, Tooze JA, Wagenknecht LE, Zhong VW, Mayer-Davis EJ. Association of Race and Ethnicity With Glycemic Control and Hemoglobin A1c Levels in Youth With Type 1 Diabetes. JAMA Netw Open. 2018 Sep 7;1(5):e181851. doi: 10.1001/jamanetworkopen.2018.1851. PMID 30370425
- [Background] Agarwal S, Hilliard M, Butler A. Disparities in Care Delivery and Outcomes in Young Adults With Diabetes. Curr Diab Rep. 2018 Jul 14;18(9):65. doi: 10.1007/s11892-018-1037-x. PMID 30008025
- [Background] Agarwal S, Kanapka LG, Raymond JK, Walker A, Gerard-Gonzalez A, Kruger D, Redondo MJ, Rickels MR, Shah VN, Butler A, Gonzalez J, Verdejo AS, Gal RL, Willi S, Long JA. Racial-Ethnic Inequity in Young Adults With Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2960-9. doi: 10.1210/clinem/dgaa236. PMID 32382736
- [Background] TODAY Study Group. Effects of metformin, metformin plus rosiglitazone, and metformin plus lifestyle on insulin sensitivity and beta-cell function in TODAY. Diabetes Care. 2013 Jun;36(6):1749-57. doi: 10.2337/dc12-2393. PMID 23704674
- [Background] Kahn SE. The relative contributions of insulin resistance and beta-cell dysfunction to the pathophysiology of Type 2 diabetes. Diabetologia. 2003 Jan;46(1):3-19. doi: 10.1007/s00125-002-1009-0. Epub 2003 Jan 11. PMID 12637977
- [Background] Gungor N, Arslanian S. Progressive beta cell failure in type 2 diabetes mellitus of youth. J Pediatr. 2004 May;144(5):656-9. doi: 10.1016/j.jpeds.2003.12.045. PMID 15127006
- [Background] Bacha F, Gungor N, Lee S, Arslanian SA. Progressive deterioration of beta-cell function in obese youth with type 2 diabetes. Pediatr Diabetes. 2013 Mar;14(2):106-11. doi: 10.1111/j.1399-5448.2012.00915.x. Epub 2012 Aug 23. PMID 22913617
- [Background] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Background] Song SH, Hardisty CA. Early onset type 2 diabetes mellitus: a harbinger for complications in later years--clinical observation from a secondary care cohort. QJM. 2009 Nov;102(11):799-806. doi: 10.1093/qjmed/hcp121. Epub 2009 Sep 4. PMID 19734298
- [Background] Sattar N, Rawshani A, Franzen S, Rawshani A, Svensson AM, Rosengren A, McGuire DK, Eliasson B, Gudbjornsdottir S. Age at Diagnosis of Type 2 Diabetes Mellitus and Associations With Cardiovascular and Mortality Risks. Circulation. 2019 May 7;139(19):2228-2237. doi: 10.1161/CIRCULATIONAHA.118.037885. PMID 30955347
- [Background] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Background] Huo X, Gao L, Guo L, Xu W, Wang W, Zhi X, Li L, Ren Y, Qi X, Sun Z, Li W, Ji Q, Ran X, Su B, Hao C, Lu J, Guo X, Zhuo H, Zhang D, Pan C, Weng J, Hu D, Yang X, Ji L. Risk of non-fatal cardiovascular diseases in early-onset versus late-onset type 2 diabetes in China: a cross-sectional study. Lancet Diabetes Endocrinol. 2016 Feb;4(2):115-24. doi: 10.1016/S2213-8587(15)00508-2. Epub 2015 Dec 17. PMID 26704379
- [Background] Dart AB, Sellers EA, Martens PJ, Rigatto C, Brownell MD, Dean HJ. High burden of kidney disease in youth-onset type 2 diabetes. Diabetes Care. 2012 Jun;35(6):1265-71. doi: 10.2337/dc11-2312. Epub 2012 Mar 19. PMID 22432116
- [Background] Brown JB, Conner C, Nichols GA. Secondary failure of metformin monotherapy in clinical practice. Diabetes Care. 2010 Mar;33(3):501-6. doi: 10.2337/dc09-1749. Epub 2009 Dec 29. PMID 20040656
- [Background] TODAY Study Group; Bjornstad P, Drews KL, Caprio S, Gubitosi-Klug R, Nathan DM, Tesfaldet B, Tryggestad J, White NH, Zeitler P. Long-Term Complications in Youth-Onset Type 2 Diabetes. N Engl J Med. 2021 Jul 29;385(5):416-426. doi: 10.1056/NEJMoa2100165. PMID 34320286
- [Background] Kim JY, Goran MI, Toledo-Corral CM, Weigensberg MJ, Shaibi GQ. Comparing glycemic indicators of prediabetes: a prospective study of obese Latino Youth. Pediatr Diabetes. 2015 Dec;16(8):640-3. doi: 10.1111/pedi.12225. Epub 2014 Nov 11. PMID 25385555
- [Background] Lawrence JM, Mayer-Davis EJ, Reynolds K, Beyer J, Pettitt DJ, D'Agostino RB Jr, Marcovina SM, Imperatore G, Hamman RF; SEARCH for Diabetes in Youth Study Group. Diabetes in Hispanic American youth: prevalence, incidence, demographics, and clinical characteristics: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2009 Mar;32 Suppl 2(Suppl 2):S123-32. doi: 10.2337/dc09-S204. PMID 19246577
- [Background] Bell RA, Mayer-Davis EJ, Beyer JW, D'Agostino RB Jr, Lawrence JM, Linder B, Liu LL, Marcovina SM, Rodriguez BL, Williams D, Dabelea D; SEARCH for Diabetes in Youth Study Group. Diabetes in non-Hispanic white youth: prevalence, incidence, and clinical characteristics: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2009 Mar;32 Suppl 2(Suppl 2):S102-11. doi: 10.2337/dc09-S202. PMID 19246575
- [Background] Sargeant JA, Brady EM, Zaccardi F, Tippins F, Webb DR, Aroda VR, Gregg EW, Khunti K, Davies MJ. Adults with early-onset type 2 diabetes (aged 18-39 years) are severely underrepresented in diabetes clinical research trials. Diabetologia. 2020 Aug;63(8):1516-1520. doi: 10.1007/s00125-020-05174-9. Epub 2020 Jun 2. PMID 32483683
- [Background] Tonnies T, Brinks R, Isom S, Dabelea D, Divers J, Mayer-Davis EJ, Lawrence JM, Pihoker C, Dolan L, Liese AD, Saydah SH, D'Agostino RB, Hoyer A, Imperatore G. Projections of Type 1 and Type 2 Diabetes Burden in the U.S. Population Aged <20 Years Through 2060: The SEARCH for Diabetes in Youth Study. Diabetes Care. 2023 Feb 1;46(2):313-320. doi: 10.2337/dc22-0945. PMID 36580405
- [Background] Lawrence JM, Divers J, Isom S, Saydah S, Imperatore G, Pihoker C, Marcovina SM, Mayer-Davis EJ, Hamman RF, Dolan L, Dabelea D, Pettitt DJ, Liese AD; SEARCH for Diabetes in Youth Study Group. Trends in Prevalence of Type 1 and Type 2 Diabetes in Children and Adolescents in the US, 2001-2017. JAMA. 2021 Aug 24;326(8):717-727. doi: 10.1001/jama.2021.11165. PMID 34427600
- [Background] Xie J, Wang M, Long Z, Ning H, Li J, Cao Y, Liao Y, Liu G, Wang F, Pan A. Global burden of type 2 diabetes in adolescents and young adults, 1990-2019: systematic analysis of the Global Burden of Disease Study 2019. BMJ. 2022 Dec 7;379:e072385. doi: 10.1136/bmj-2022-072385. PMID 36740855
- [Background] Wu H, Patterson CC, Zhang X, Ghani RBA, Magliano DJ, Boyko EJ, Ogle GD, Luk AOY. Worldwide estimates of incidence of type 2 diabetes in children and adolescents in 2021. Diabetes Res Clin Pract. 2022 Mar;185:109785. doi: 10.1016/j.diabres.2022.109785. Epub 2022 Feb 18. PMID 35189261
- [Background] Perng W, Conway R, Mayer-Davis E, Dabelea D. Youth-Onset Type 2 Diabetes: The Epidemiology of an Awakening Epidemic. Diabetes Care. 2023 Mar 1;46(3):490-499. doi: 10.2337/dci22-0046. PMID 36812420
- [Background] Falkner B, Gidding S. Life-Course Implications of Pediatric Risk Factors for Cardiovascular Disease. Can J Cardiol. 2021 May;37(5):766-775. doi: 10.1016/j.cjca.2021.02.001. Epub 2021 Feb 11. PMID 33581191
- [Background] American Diabetes Association Professional Practice Committee. 4. Comprehensive Medical Evaluation and Assessment of Comorbidities: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S52-S76. doi: 10.2337/dc24-S004. PMID 38078591
- [Background] American Diabetes Association Professional Practice Committee. 14. Children and Adolescents: Standards of Care in Diabetes-2024. Diabetes Care. 2024 Jan 1;47(Suppl 1):S258-S281. doi: 10.2337/dc24-S014. PMID 38078582
- [Background] Misra A. Ethnic-Specific Criteria for Classification of Body Mass Index: A Perspective for Asian Indians and American Diabetes Association Position Statement. Diabetes Technol Ther. 2015 Sep;17(9):667-71. doi: 10.1089/dia.2015.0007. Epub 2015 Apr 22. PMID 25902357
- [Background] Florido R, Daya NR, Ndumele CE, Koton S, Russell SD, Prizment A, Blumenthal RS, Matsushita K, Mok Y, Felix AS, Coresh J, Joshu CE, Platz EA, Selvin E. Cardiovascular Disease Risk Among Cancer Survivors: The Atherosclerosis Risk In Communities (ARIC) Study. J Am Coll Cardiol. 2022 Jul 5;80(1):22-32. doi: 10.1016/j.jacc.2022.04.042. PMID 35772913
- [Background] Triant VA, Lee H, Hadigan C, Grinspoon SK. Increased acute myocardial infarction rates and cardiovascular risk factors among patients with human immunodeficiency virus disease. J Clin Endocrinol Metab. 2007 Jul;92(7):2506-12. doi: 10.1210/jc.2006-2190. Epub 2007 Apr 24. PMID 17456578
- [Background] Freiberg MS, Chang CC, Kuller LH, Skanderson M, Lowy E, Kraemer KL, Butt AA, Bidwell Goetz M, Leaf D, Oursler KA, Rimland D, Rodriguez Barradas M, Brown S, Gibert C, McGinnis K, Crothers K, Sico J, Crane H, Warner A, Gottlieb S, Gottdiener J, Tracy RP, Budoff M, Watson C, Armah KA, Doebler D, Bryant K, Justice AC. HIV infection and the risk of acute myocardial infarction. JAMA Intern Med. 2013 Apr 22;173(8):614-22. doi: 10.1001/jamainternmed.2013.3728. PMID 23459863
- [Background] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Background] Frost F, Nazareth D, Fauchier L, Wat D, Shelley J, Austin P, Walshaw MJ, Lip GYH. Prevalence, risk factors and outcomes of cardiac disease in cystic fibrosis: a multinational retrospective cohort study. Eur Respir J. 2023 Oct 26;62(4):2300174. doi: 10.1183/13993003.00174-2023. Print 2023 Oct. PMID 37474158
- [Background] Sandouk Z, Nachawi N, Simon R, Wyckoff J, Putman MS, Kiel S, Soltman S, Moran A, Moheet A. Coronary artery disease in patients with cystic fibrosis - A case series and review of the literature. J Clin Transl Endocrinol. 2022 Oct 5;30:100308. doi: 10.1016/j.jcte.2022.100308. eCollection 2022 Dec. PMID 36267108
- [Background] Roberts R, Speight L, Lee J, George L, Ketchell RI, Lau D, Duckers J. Retinal screening of patients with cystic fibrosis-related diabetes in Wales -- a real eye opener. J Cyst Fibros. 2015 Mar;14(2):282-4. doi: 10.1016/j.jcf.2014.07.014. Epub 2014 Sep 13. PMID 25224328
- [Background] Lind-Ayres M, Thomas W, Holme B, Mauer M, Caramori ML, Moran A. Microalbuminuria in patients with cystic fibrosis. Diabetes Care. 2011 Jul;34(7):1526-8. doi: 10.2337/dc10-2231. Epub 2011 May 11. PMID 21562324
- [Background] Schwarzenberg SJ, Thomas W, Olsen TW, Grover T, Walk D, Milla C, Moran A. Microvascular complications in cystic fibrosis-related diabetes. Diabetes Care. 2007 May;30(5):1056-61. doi: 10.2337/dc06-1576. Epub 2007 Feb 23. PMID 17322485
- [Background] Colomba J, Boudreau V, Lehoux-Dubois C, Desjardins K, Coriati A, Tremblay F, Rabasa-Lhoret R. The main mechanism associated with progression of glucose intolerance in older patients with cystic fibrosis is insulin resistance and not reduced insulin secretion capacity. J Cyst Fibros. 2019 Jul;18(4):551-556. doi: 10.1016/j.jcf.2019.01.009. Epub 2019 Jan 30. PMID 30711385
- [Background] Blackman SM, Hsu S, Vanscoy LL, Collaco JM, Ritter SE, Naughton K, Cutting GR. Genetic modifiers play a substantial role in diabetes complicating cystic fibrosis. J Clin Endocrinol Metab. 2009 Apr;94(4):1302-9. doi: 10.1210/jc.2008-2186. Epub 2009 Jan 6. PMID 19126627
- [Background] Blackman SM, Hsu S, Ritter SE, Naughton KM, Wright FA, Drumm ML, Knowles MR, Cutting GR. A susceptibility gene for type 2 diabetes confers substantial risk for diabetes complicating cystic fibrosis. Diabetologia. 2009 Sep;52(9):1858-65. doi: 10.1007/s00125-009-1436-2. Epub 2009 Jul 8. PMID 19585101
- [Background] Blackman SM, Commander CW, Watson C, Arcara KM, Strug LJ, Stonebraker JR, Wright FA, Rommens JM, Sun L, Pace RG, Norris SA, Durie PR, Drumm ML, Knowles MR, Cutting GR. Genetic modifiers of cystic fibrosis-related diabetes. Diabetes. 2013 Oct;62(10):3627-35. doi: 10.2337/db13-0510. Epub 2013 May 13. PMID 23670970
- [Background] Aksit MA, Pace RG, Vecchio-Pagan B, Ling H, Rommens JM, Boelle PY, Guillot L, Raraigh KS, Pugh E, Zhang P, Strug LJ, Drumm ML, Knowles MR, Cutting GR, Corvol H, Blackman SM. Genetic Modifiers of Cystic Fibrosis-Related Diabetes Have Extensive Overlap With Type 2 Diabetes and Related Traits. J Clin Endocrinol Metab. 2020 May 1;105(5):1401-15. doi: 10.1210/clinem/dgz102. PMID 31697830
- [Background] Malik SS, Padmanabhan D, Hull-Meichle RL. Pancreas and islet morphology in cystic fibrosis: clues to the etiology of cystic fibrosis-related diabetes. Front Endocrinol (Lausanne). 2023 Nov 23;14:1269139. doi: 10.3389/fendo.2023.1269139. eCollection 2023. PMID 38075070
- [Background] Norris AW, Ode KL, Merjaneh L, Sanda S, Yi Y, Sun X, Engelhardt JF, Hull RL. Survival in a bad neighborhood: pancreatic islets in cystic fibrosis. J Endocrinol. 2019 Apr;241(1):R35-R50. doi: 10.1530/JOE-18-0468. PMID 30759072
- [Background] Sheikh S, Gudipaty L, De Leon DD, Hadjiliadis D, Kubrak C, Rosenfeld NK, Nyirjesy SC, Peleckis AJ, Malik S, Stefanovski D, Cuchel M, Rubenstein RC, Kelly A, Rickels MR. Reduced beta-Cell Secretory Capacity in Pancreatic-Insufficient, but Not Pancreatic-Sufficient, Cystic Fibrosis Despite Normal Glucose Tolerance. Diabetes. 2017 Jan;66(1):134-144. doi: 10.2337/db16-0394. Epub 2016 Aug 5. PMID 27495225
- [Background] Nyirjesy SC, Sheikh S, Hadjiliadis D, De Leon DD, Peleckis AJ, Eiel JN, Kubrak C, Stefanovski D, Rubenstein RC, Rickels MR, Kelly A. beta-Cell secretory defects are present in pancreatic insufficient cystic fibrosis with 1-hour oral glucose tolerance test glucose >/=155 mg/dL. Pediatr Diabetes. 2018 Nov;19(7):1173-1182. doi: 10.1111/pedi.12700. Epub 2018 Jun 21. PMID 29885044
- [Background] Moheet A, Moran A. New Concepts in the Pathogenesis of Cystic Fibrosis-Related Diabetes. J Clin Endocrinol Metab. 2022 May 17;107(6):1503-1509. doi: 10.1210/clinem/dgac020. PMID 35106591
- [Background] Szentpetery S, Fernandez GS, Schechter MS, Jain R, Flume PA, Fink AK. Obesity in Cystic fibrosis: prevalence, trends and associated factors data from the US cystic fibrosis foundation patient registry. J Cyst Fibros. 2022 Sep;21(5):777-783. doi: 10.1016/j.jcf.2022.03.010. Epub 2022 Apr 5. PMID 35396178
- [Background] Harindhanavudhi T, Wang Q, Dunitz J, Moran A, Moheet A. Prevalence and factors associated with overweight and obesity in adults with cystic fibrosis: A single-center analysis. J Cyst Fibros. 2020 Jan;19(1):139-145. doi: 10.1016/j.jcf.2019.10.004. Epub 2019 Nov 11. PMID 31727452
- [Background] Sawicki GS, McKone EF, Pasta DJ, Millar SJ, Wagener JS, Johnson CA, Konstan MW. Sustained Benefit from ivacaftor demonstrated by combining clinical trial and cystic fibrosis patient registry data. Am J Respir Crit Care Med. 2015 Oct 1;192(7):836-42. doi: 10.1164/rccm.201503-0578OC. PMID 26132840
- [Background] Rowe SM, McColley SA, Rietschel E, Li X, Bell SC, Konstan MW, Marigowda G, Waltz D, Boyle MP; VX09-809-102 Study Group. Lumacaftor/Ivacaftor Treatment of Patients with Cystic Fibrosis Heterozygous for F508del-CFTR. Ann Am Thorac Soc. 2017 Feb;14(2):213-219. doi: 10.1513/AnnalsATS.201609-689OC. PMID 27898234
- [Background] Rowe SM, Daines C, Ringshausen FC, Kerem E, Wilson J, Tullis E, Nair N, Simard C, Han L, Ingenito EP, McKee C, Lekstrom-Himes J, Davies JC. Tezacaftor-Ivacaftor in Residual-Function Heterozygotes with Cystic Fibrosis. N Engl J Med. 2017 Nov 23;377(21):2024-2035. doi: 10.1056/NEJMoa1709847. Epub 2017 Nov 3. PMID 29099333
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Background] Nichols DP, Paynter AC, Heltshe SL, Donaldson SH, Frederick CA, Freedman SD, Gelfond D, Hoffman LR, Kelly A, Narkewicz MR, Pittman JE, Ratjen F, Rosenfeld M, Sagel SD, Schwarzenberg SJ, Singh PK, Solomon GM, Stalvey MS, Clancy JP, Kirby S, Van Dalfsen JM, Kloster MH, Rowe SM; PROMISE Study group. Clinical Effectiveness of Elexacaftor/Tezacaftor/Ivacaftor in People with Cystic Fibrosis: A Clinical Trial. Am J Respir Crit Care Med. 2022 Mar 1;205(5):529-539. doi: 10.1164/rccm.202108-1986OC. PMID 34784492
- [Background] Middleton PG, Mall MA, Drevinek P, Lands LC, McKone EF, Polineni D, Ramsey BW, Taylor-Cousar JL, Tullis E, Vermeulen F, Marigowda G, McKee CM, Moskowitz SM, Nair N, Savage J, Simard C, Tian S, Waltz D, Xuan F, Rowe SM, Jain R; VX17-445-102 Study Group. Elexacaftor-Tezacaftor-Ivacaftor for Cystic Fibrosis with a Single Phe508del Allele. N Engl J Med. 2019 Nov 7;381(19):1809-1819. doi: 10.1056/NEJMoa1908639. Epub 2019 Oct 31. PMID 31697873
- [Background] Heijerman HGM, McKone EF, Downey DG, Van Braeckel E, Rowe SM, Tullis E, Mall MA, Welter JJ, Ramsey BW, McKee CM, Marigowda G, Moskowitz SM, Waltz D, Sosnay PR, Simard C, Ahluwalia N, Xuan F, Zhang Y, Taylor-Cousar JL, McCoy KS; VX17-445-103 Trial Group. Efficacy and safety of the elexacaftor plus tezacaftor plus ivacaftor combination regimen in people with cystic fibrosis homozygous for the F508del mutation: a double-blind, randomised, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1940-1948. doi: 10.1016/S0140-6736(19)32597-8. Epub 2019 Oct 31. PMID 31679946
- [Background] Davies JC, Wainwright CE, Canny GJ, Chilvers MA, Howenstine MS, Munck A, Mainz JG, Rodriguez S, Li H, Yen K, Ordonez CL, Ahrens R; VX08-770-103 (ENVISION) Study Group. Efficacy and safety of ivacaftor in patients aged 6 to 11 years with cystic fibrosis with a G551D mutation. Am J Respir Crit Care Med. 2013 Jun 1;187(11):1219-25. doi: 10.1164/rccm.201301-0153OC. PMID 23590265